CLINICAL TRIAL: NCT03806972
Title: Short and Long Term Prognosis of Patients Admitted to the Emergency Department With Acute Heart Failure
Brief Title: Short and Long Term Prognosis of Patients Admitted to the ED With Acute Heart Failure
Acronym: CRF
Status: Recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: CRF
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Heart failure (HF) is the leading cause of hospitalization ,rehospitalization and mortality for adults over 65 years of age.

This study aimed to assess mortality, and hospitalization rates at 30 days and one year after dicharge of patients with heart failure (HF) with reduced ejection fraction (HFrEF) compared to HF with preserved ejection fraction (HFpEF).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the ED of Monastir with a principal discharge diagnosis code for HF.

Exclusion Criteria:

* Pregnant or breast feeding women. Alteration of consciousness GCS < 15 Critically ill patients needing immediate mechanical hemodynamic of ventilatory support.

Inability to follow instructions or comply with follow-up procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included all patients ,with either reduced ejection fraction (HFrEF) defined as LVEF <45% or preserved ejection fraction (HFpEF) defined as LVEF ≥45% ,admitted to the ED of Monastir from 2009 with a principal discharge diagnosis code for HF. The diagnosis of HF categories should rely on the recent transthoracic echocardiographic findings and clinical judgement according to the guidelines.Collected data include clinical features biological markers (BNP or NTpro BNP) and echocardiography findings. The diagnosis of HF categories should rely on the recent transthoracic echocardiographic findings and clinical judgement according to the guidelines. A follow-up period of at least 1 year was required to notice all cause mortality and preferably HF-specific rehospitalization .
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-06-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Death or readmission rates | within 365 days after hospital discharge
  A composite outcome of Death or readmission within 365 days of hospital discharge

SECONDARY OUTCOMES:
Death or readmission rates | within 30 days after hospital discharge
  A composite outcome of Death or readmission within 30 days of hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — university Hospital of Monastir
Locations (1):
- Emergency Departement, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castello LM, Molinari L, Renghi A, Peruzzi E, Capponi A, Avanzi GC, Pirisi M. Acute decompensated heart failure in the emergency department: Identification of early predictors of outcome. Medicine (Baltimore). 2017 Jul;96(27):e7401. doi: 10.1097/MD.0000000000007401. PMID 28682895
- [Background] Searle J, Frick J, Mockel M. Acute heart failure facts and numbers: acute heart failure populations. ESC Heart Fail. 2016 Jun;3(2):65-70. doi: 10.1002/ehf2.12092. Epub 2016 Apr 25. PMID 27818780